CLINICAL TRIAL: NCT01813903
Title: Family Welfare Pilot Intervention Study at Finnish Welfare Clinics
Brief Title: Family Welfare Pilot Intervention Study
Acronym: HYPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Tampere University (Other); University of Helsinki (Other); University of Jyvaskyla (Other); VTT Technical Research Centre of Finland (Other); The Finnish Heart Association (Unknown); The National Consumer Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THL10433
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nutrition (Experimental): Intensified dietary counseling and use of web application.
  Interventions: Behavioral: Intensified dietary counseling
- Flexible mind (Experimental): Use of mobile applications.
  Interventions: Behavioral: Mobile application
- Normal maternity clinic visits (No Intervention): In control maternity clinics, nurses continue their usual counseling.

INTERVENTIONS:
Behavioral: Intensified dietary counseling — The intervention is completed by public health nurses who will be trained to provide family-centered empowering and motivational lifestyle counseling at the normal health check visit. Parents expecting child will use web application developed for nutritional counseling. Web application consists of dietary questionnaire from which the parents will receive immediately automatic feedback. Feedback concerns the quality of diet in relation to the Finnish nutrition recommendations. Feedback will be given in an encouraging format. Own targets of food changes can also be recorded in the application, and the application can be used to monitor how they are achieved.
  Arms: Nutrition
Behavioral: Mobile application — Mothers expecting child will use mobile application. Mobile application consists of text, audio and video exercises, which are aimed to increase the psychological flexibility and thus mental and physical well-being.
  Arms: Flexible mind

SUMMARY:
The purpose of this study was to test internet and mobile-based applications to support motivating lifestyle counseling to promote healthy eating habits of the mothers and their spouses expecting first child. The feasibility of the intervention will be evaluated in the pilot.

DETAILED DESCRIPTION:
Lifestyle habits during pregnancy have long-term effects of baby's as well as mother's health. Pregnancy period is a favorable time for lifestyle changes, as the parents usually have motivation and assets to change lifestyle. Maternity welfare clinic is the place to promote healthy lifestyles because most Finnish families expecting child visit there at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* All families expecting their child at their standard 8-10 pregnancy weeks welfare clinic visit

Exclusion Criteria:

* Parents are under 18-year-old
* Parents do not speak Finnish
* Parents do not have internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Food consumption of the parents | 7 months
  Measured with Food Frequency Questionnaire
Maternal post-natal depression | 9 months
  Measured with Edinburgh Postnatal Depression Scale (EDPS)

SECONDARY OUTCOMES:
Food and health related attitudes and aims of the parent's | 9 months
  Questions about food and health related attitudes and aims
Psychological flexibility of the parent's | 9 months
  Measured with Acceptance & Action Questionnaire (AAQ-2)
Mental health of the parent's | 9 months
  Measured with Mental Health Continuum Short Form (MHC-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Suvi I Virtanen, Professor, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- Maternal welfare clinics, Vantaa, Finland